CLINICAL TRIAL: NCT04804956
Title: Mesorectal Microbiome as a Prognostic Factor in Patients With Rectal Cancer and Analysis of it's Applicability in Neoadjuvant Treatment
Brief Title: Mesorectal Microbiome as a Prognostic Factor in Patients With Rectal Cancer
Acronym: BIORECTUM
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Girona Dr. Josep Trueta (Network)
Collaborators: Girona Biomedical Research Institute (Unknown)
Responsible Party: Principal Investigator, Antoni Codina Cazador, PhD, MD, Principal Investigator, University Hospital of Girona Dr. Josep Trueta
Other Study IDs: 2012.028
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Rectal Cancer
Keywords: Rectal Neoplasms; Colorectal surgery; Gastrointestinal Microbiome
MeSH Terms: conditions — Rectal Neoplasms | interventions — Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, faeces, rectal mucosa, mesorectal, subcutaneous and visceral adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early-rectal cancer: The patients to be included in this group will be those with Stage I (initial tumor stage). The tumors classified in stage I will be tumors in which the invasion of the submucosa and / or the invasion of the muscularis propria occur. This group will include patients diagnosed preoperatively with tumor stage T1-T2 N0.
  Interventions: Procedure: Stool sample; Procedure: Rectal mucosa sample; Procedure: Mesorectal adipose tissue sample; Procedure: Subcutaneous adipose tissue sample; Procedure: Visceral adipose tissue sample; Behavioral: Dietary assessment
- Advanced-rectal cancer: The patients to be included in this group will be those with Stages II and III, that is, advanced tumors at the time of preoperative diagnosis. Tumors included in this group invade the perirectal fat and / or the surface of the visceral peritoneum and / or invade or adhere to adjacent organs or structures. In addition, any tumor stage with lymph nodes without distant metastases will be included in this group.
  Interventions: Procedure: Stool sample; Procedure: Rectal mucosa sample; Procedure: Mesorectal adipose tissue sample; Procedure: Subcutaneous adipose tissue sample; Procedure: Visceral adipose tissue sample; Behavioral: Dietary assessment
- Synchronous metastasis -rectal cancer: The patients to be included in this group will be those with Stage IV (disseminated tumor stage) in the initial study of the disease. Patients with distant metastases in one organ or more than one organ will be included.
  Interventions: Procedure: Stool sample; Procedure: Rectal mucosa sample; Procedure: Mesorectal adipose tissue sample; Procedure: Subcutaneous adipose tissue sample; Procedure: Visceral adipose tissue sample; Behavioral: Dietary assessment

INTERVENTIONS:
Procedure: Stool sample — One stool sample will be taken at baseline for microbiota characterization
Procedure: Rectal mucosa sample — Characterization of tissue microbiota before and after surgery.
Procedure: Mesorectal adipose tissue sample — Characterization of tissue microbiota and dysfunction
Procedure: Subcutaneous adipose tissue sample — Characterization of tissue microbiota and dysfunction
Procedure: Visceral adipose tissue sample — Characterization of tissue microbiota and dysfunction
Behavioral: Dietary assessment — Dietary assessment will be taken at baseline

SUMMARY:
The equilibrium of intestinal microorganisms is essential for health an imbalance has been associated with an increased risk in the development of different pathologies; including colorectal cancer.

Rectal cancer is the third most common neoplasm worldwide and the complete excision of the mesorectum is a major prognostic factor.

The identification of microorganisms in the adipose tissue that surrounds the small intestine in inflammatory diseases, together with bacterial alterations found in colonic mucosa and feces in patients with rectal cancer in comparison with healthy individuals indicates that microbiome alteration plays an essential role in pathogenesis.

The mesorectal microbiome in rectal cancer patients stills unknown and given its importance in the prognostic of the disease the goal of this study is to identify microbial profiles that allow predicting rectal cancer patients with a poor prognosis.

DETAILED DESCRIPTION:
The 5-year survival rate for patients with rectal cancer is 64%. Despite the development of personalized cancer treatments, the implantation of surgical approaches with more precise fields of vision and the current prognostic factors based on the quality of resection of the surgical specimen (intact margins and complete resection of the mesorectum), the long-term results for patients with rectal cancer remain grim.

Recently, it has been shown that dysfunctional fat tissue is characterized by tissue remodeling, grater lipids deposits and high adipokines secretion generates a pro inflammatory state, hypoxia and angiogenesis. These products generated by dysfunctional peritumoral adipose tissue create an ideal microenvironment for initiation and tumor progression.

The presence of microbiome in the mesentery of patients with colitis has confirmed the translocation of microorganisms from the intestine to adjacent tissues, together with the differences found in the bacterial composition in colonic mucosa and fecal samples between patients with rectal cancer and healthy individuals, and the prognosis value of the quality of mesorectum resection suggests that the microbiome present in lymph-fatty tissue in patients with rectal cancer may be a key element in mesorectum dysfunction, progression and dissemination of oncological disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer that will undergo anterior resection for rectal cancer.
* Age ≥ 18 years
* Histology proven adenocarcinoma or adenoma with or without chemotherapy or neoadjuvant radiochemotherapy
* Tumoral stage equal or grater than T1
* Attempt to R0 resection
* Signed informed consent by the patient and by the researcher
* Dietary Questionnaire completed

Exclusion Criteria:

* Colorectal tumor with different histology to adenocarcinoma or adenoma
* History of colorectal cancer surgery different to the local excision
* Patients with psychiatric illness, addiction or disorder with inability to understand informed consent
* Inability to read or understand any of the languages of the informed consent and questionnaires (Catalan, spanish)
* Another synchronous malignancy
* Emergency Surgery
* Any patient that medical characteristics present an individual risk raised to be included and complete the study
* Severe kidney or liver disease
* Systemic disease with inflammatory activity, such as rheumatoid arthritis, Crohn's disease, asthma, chronic infection (HIV,TBC).
* Pregnancy and lactation
* Severe disorder of eating behaviour
* Clinical symptoms and sings of infection in the previous month
* Antibiotic, antifungal and antiviral treatment for the last 3 months
* Anti-inflammatory chronic treatment
* Major psychiatric antecedents
* Excessive alcohol intake or drug abuse

Ages: 18 Years to 18 Years | Sex: All
Age Groups: Adult
Study Population: Patients diagnosed with rectal cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Identification of mesorectal microbial biomarkers as prognostic factor for rectal cancer | Up to 5 years after rectal cancer surgery
  Correlation between mesorectal microbial signatures and survival

SECONDARY OUTCOMES:
Mesorectal microbiome evaluation | Up to 1 month after rectal cancer surgery
  Qualitative and quantitative analysis of the mesorectal microbiome in patients with rectal cancer
Evaluation of mesorectal dysfunctionality and its correlation with microbial dysbiosis | Up to 1 month after rectal cancer surgery
  Analysis of mesorectal tissue inflammation, angiogenesis and hypoxia and its correlation with microbial dysbiosis
Evaluation of mesorectal dysfunctionality and dysbiosis on tumor progression | Up to 1 month after rectal cancer surgery
  Correlation between mesorectal dysfunction and response to neoadjuvant treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Dr. Josep Trueta de Girona, Girona, Spain